CLINICAL TRIAL: NCT05666362
Title: Hemodynamic Response Of Premature Brain To Pain During Retinopathy Of Prematurity Screening: A Randomized Controlled Trial
Brief Title: Hemodynamic Response to Pain During Retinopathy Of Prematurity Screening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107389
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Preterm
MeSH Terms: conditions — Premature Birth | interventions — benoxinate; Population Groups; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : ( benoxinate hydrochloride 0.4% group ) (Active Comparator): They will receive benoxinate hydrochloride 0.4% immediately before fundus examination .
  Interventions: Drug: benoxinate hydrochloride 0.4% group
- Group 2 : ( control group ) (Placebo Comparator): They will receive saline drops instead of benoxinate hydrochloride 0.4%. Randomization: simple randomization sampling using sealed envelope technique.
  Interventions: Drug: saline 0.9% .

INTERVENTIONS:
Drug: benoxinate hydrochloride 0.4% group — They will receive benoxinate hydrochloride 0.4% immediately before fundus
  Arms: Group 1 : ( benoxinate hydrochloride 0.4% group )
Drug: saline 0.9% . — They will receive saline 0.9% before fundus examination in each eye .
  Arms: Group 2 : ( control group )

SUMMARY:
Study of cerebral hemodynamic changes in preterm infant and the effect of topical anesthetic eye drops ( benoxinate hydrochloride 0.4% ) on PIPP score and cerebral hemodynamic changes during fundus examination in neonates with gestational age ≤ 34 weeks or birth weight ≤ 2.000 Kg regardless their gestational age , after postnatal day 28.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants with gestational age ≤34 weeks or infant with birth weight ≤ 2.000 Kg regardless their gestational age,with postnatal age ≥ 28 days undergoing routine ROP screening.

Exclusion Criteria:

Patients with any of the following will be excluded at the time of assessment:

* Evidence of intrauterine infection (TORCH).
* Chromosomal abnormalities.
* Major congenital anomalies.
* Major brain pathology such as Grade 3-4 intraventricular hemorrhage and periventricular leukomalacia.

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
1-Clinical assessment: | 28 days postnatal age (time of screen of retinopathy of prematurity ,ROP)
  Pain score will be evaluated by using the premature infant pain profile (PIPP) assessed by the caring bedside nurse during fundus examination. It consists of heart rate(beat/minute), peripheral oxygen saturation in the right hand(%), and mean arterial blood pressure (mmHg).
2-Near-infrared spectroscopy (NIRS): | 28 days postnatal age (time of screen of retinopathy of prematurity ,ROP)
  Measurements of cerebral oxygenation (crSO2) in (%) will be done by using near infrared spectroscopy (NIRS), device (INVOSTM 5100C Cerebral/ Somatic Oximeter Monitor; Covidien) by placing a neonatal brain sensor on the right frontoparietal area of the scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa Hafez, MBChB, Principal Investigator — Faculty of medicine, Alexandria University, Egypt; Hesham Ghazal, PhD, Study Director — Faculty of medicine, Alexandria University, Egypt
Locations (1):
- Marwa Mohamed Farag, Alexandria, Egypt